CLINICAL TRIAL: NCT06586372
Title: CRP,CRP/Alb Ratio, N/L Ratio in Predictors of Both Systemic Infection and Survival in Patient with Sepsis
Brief Title: CRP,CRP/Alb Ratio, N/L Ratio in Predictors of Both Systemic Infection and Survival in Patient with Sepsis in Assiut University Hospitals
Status: Not yet recruiting | Type: Observational
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Esraa Ahmed Mohamed Gomaa, doctor, Assiut University
Other Study IDs: predictors /Survival /sepsis
Record Dates: First submitted 2024-09-04; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Sepsis; Systemic Infection
MeSH Terms: conditions — Sepsis; Toxemia

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
the goal of this study is to asses the value of biomarker (CRP, CRP/Alb ratio, N/L ratio) in predictor of the outcome in normotensive patients with sepsis.

The main question it aims to answer is:

Does biomarker (CRP, CRP/Alb ratio, N/L ratio) can predict the outcome in patients with sepsis ?

DETAILED DESCRIPTION:
Sepsis is an unusual systemic reaction to what is sometimes an otherwise ordinary infection, and it probably represents a pattern of response by the immune system to injury. A hyper-inflammatory response is followed by an immunosuppressive phase during which multiple organ dysfunction is present and the patient is susceptible to nosocomial infection.

A biomarker describes a measurable indicator of a patient's clinical condition that can be measured accurately and reproducibly. Biomarkers offer utility for diagnosis, prognosis, early disease recognition, risk stratification, appropriate treatment (theranostics), and trial enrichment for patients with sepsis or suspected sepsis C-reactive protein (CRP) is an acute-phase protein that is produced following stimulation by various cytokines in response to infection, ischemia, trauma, and other inflammatory conditions . High CRP levels have been studied in relation to prognosis and mortality in critically ill patients . On the other hand, low serum albumin is known to be associated with poor prognosis and mortality . Based on this knowledge, we speculated that the ratio of CRP to albumin could be used as a predictive marker for mortality.

Recently, the CRP/albumin ratio, a combination of markers for systemic inflammation and nutritional status, has been extensively studied as an independent prognostic marker in patients with infection, malignancy, and other diseases . However, there are relatively few studies conducted focusing on critical care patients in the ICU Among the plethora of biomarkers available to clinicians investigating septic patients in the Emergency Department (ED), white blood cell count (WBC) are always taken into consideration due to their availability and low cost. Serial measurement of RP, is useful for clinicians' decision-making, as its serum levels correlate with the syndrome evo-lution .Neutrophil-to-lymphocyte ratio (NLR) calculated from the complete blood count seems to be a reasonable tool for assessment during the sepsis course (8, 9).

ELIGIBILITY:
Inclusion Criteria:

* Patients with sepsis with normal blood pressure

Exclusion Criteria:

* 1) Patients with history of corticosteroid therapy or antibiotic use before admission.

  2) Patients with hematologic disorders, malignant diseases, chemotherapy or radiotherapy within the previous month .

  3)Patients with shock

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: the patients will be diagnosed according to international criteria and sepsis-3 definitions
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2024-10-01 (Estimated); Primary Completion 2025-10-30 (Estimated); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
CRP level in patients with sepsis | baseline
CRP/Alb ratio level in patients with sepsis | baseline

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kinoshita A, Onoda H, Imai N, Iwaku A, Oishi M, Tanaka K, Fushiya N, Koike K, Nishino H, Matsushima M. The C-reactive protein/albumin ratio, a novel inflammation-based prognostic score, predicts outcomes in patients with hepatocellular carcinoma. Ann Surg Oncol. 2015 Mar;22(3):803-10. doi: 10.1245/s10434-014-4048-0. Epub 2014 Sep 5. PMID 25190127
- [Background] Saito H, Kono Y, Murakami Y, Shishido Y, Kuroda H, Matsunaga T, Fukumoto Y, Osaki T, Ashida K, Fujiwara Y. Prognostic Significance of the Preoperative Ratio of C-Reactive Protein to Albumin and Neutrophil-Lymphocyte Ratio in Gastric Cancer Patients. World J Surg. 2018 Jun;42(6):1819-1825. doi: 10.1007/s00268-017-4400-1. PMID 29270656
- [Background] Ranzani OT, Zampieri FG, Forte DN, Azevedo LC, Park M. C-reactive protein/albumin ratio predicts 90-day mortality of septic patients. PLoS One. 2013;8(3):e59321. doi: 10.1371/journal.pone.0059321. Epub 2013 Mar 12. PMID 23555017
- [Background] Artero A, Zaragoza R, Camarena JJ, Sancho S, Gonzalez R, Nogueira JM. Prognostic factors of mortality in patients with community-acquired bloodstream infection with severe sepsis and septic shock. J Crit Care. 2010 Jun;25(2):276-81. doi: 10.1016/j.jcrc.2009.12.004. Epub 2010 Feb 10. PMID 20149587
- [Background] Lobo SM, Lobo FR, Bota DP, Lopes-Ferreira F, Soliman HM, Melot C, Vincent JL. C-reactive protein levels correlate with mortality and organ failure in critically ill patients. Chest. 2003 Jun;123(6):2043-9. doi: 10.1378/chest.123.6.2043. PMID 12796187
- [Background] Villacorta H, Masetto AC, Mesquita ET. C-reactive protein: an inflammatory marker with prognostic value in patients with decompensated heart failure. Arq Bras Cardiol. 2007 May;88(5):585-9. doi: 10.1590/s0066-782x2007000500014. English, Portuguese. PMID 17589635
- [Background] Ho KM, Dobb GJ, Lee KY, Towler SC, Webb SA. C-reactive protein concentration as a predictor of intensive care unit readmission: a nested case-control study. J Crit Care. 2006 Sep;21(3):259-65. doi: 10.1016/j.jcrc.2006.01.005. PMID 16990094
- [Background] Thijs LG, Hack CE. Time course of cytokine levels in sepsis. Intensive Care Med. 1995 Nov;21 Suppl 2:S258-63. doi: 10.1007/BF01740764. PMID 8636533
- [Background] Barichello T, Generoso JS, Singer M, Dal-Pizzol F. Biomarkers for sepsis: more than just fever and leukocytosis-a narrative review. Crit Care. 2022 Jan 6;26(1):14. doi: 10.1186/s13054-021-03862-5. PMID 34991675
- [Background] Faix JD. Biomarkers of sepsis. Crit Rev Clin Lab Sci. 2013 Jan-Feb;50(1):23-36. doi: 10.3109/10408363.2013.764490. PMID 23480440
- [Background] Rello J, Valenzuela-Sanchez F, Ruiz-Rodriguez M, Moyano S. Sepsis: A Review of Advances in Management. Adv Ther. 2017 Nov;34(11):2393-2411. doi: 10.1007/s12325-017-0622-8. Epub 2017 Oct 11. PMID 29022217